CLINICAL TRIAL: NCT01946022
Title: In Vitro Evaluation of Luteinized Granulosa Cells After Being Submitted to in Vitro Fertilization Protocols With Gonadotropin-Releasing Hormone (GnRH) Agonist and GnRH Antagonist
Brief Title: Evaluation of Granulosa Cells Function After IVF Protocols
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 13-0120; HCPA (Other: Hospital de Clínicas de Porto Alegre)
Record Dates: First submitted 2013-08-02; First posted 2013-09-19 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-11

CONDITIONS: Infertility; In Vitro Fertilization Protocols
Keywords: infertility; ovulation induction; luteal phase; granulosa cells function; GnRH agonist and antagonist; HMG; FSHr
MeSH Terms: conditions — Infertility

ARMS (2):
- GnRH Agonist (Active Comparator): GnRH long agonist protocol of invitro fertilization
  Interventions: Drug: randomization between the two GnRH analogues (agonist and antagonist)
- GnRH Antagonist (Active Comparator): GnRH fixed antagonist protocol of in vitro fertilization
  Interventions: Drug: randomization between the two GnRH analogues (agonist and antagonist)

INTERVENTIONS:
Drug: randomization between the two GnRH analogues (agonist and antagonist)

SUMMARY:
This study is intended to evaluate ovarian cells after being submitted do different in vitro fertilization protocols. The investigators will analyze hormones secretion and intracellular mechanisms of these cells comparing the GnRH agonist protocol and the GnRH antagonist protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patient age limit: 39 years
* Follicle Stimulating Hormone (FSH) < 10 micrometer (mU) / Liter
* Antral follicular count > 12
* Regular menses (25 to 35 days)
* More than 3 oocytes after ovarian punction
* Anti Mullerian between 1 e 3 ng/ml

Exclusion Criteria:

* Patients submitted to intracytoplasmatic sperm injection (ICSI)
* Ovarian mass or cyst
* Clinical / endocrine pathologies

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Evaluation of steroid secretion and enzyme expression in in vitro luteinized granulosa cells | after 48h in media culture
  evaluation of granulosa cells hormone secretion and enzyme expression in media culture 48 hours after ovarian punction
Number of retrieved oocytes | After the ovarian punction
  Immediately after the ovarian punction the number of retrieved oocytes will be evaluated

SECONDARY OUTCOMES:
number of embryos | 3 to 5 days after ovarian punction
  the embryologist will verify the number of embryos after 3 to 5 days from the ovarian punction
Subgroup analyses comparing FSH versus HMG protocols | after ovarian punction
  It will be verified the differences between the two types of gonadotrophins in ovarian stimulation regarding: units of gonadotrophins used, number of retrieved oocytes,number of embryos and embryo score

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Projeto Cegonha, Porto Alegre, Rio Grande do Sul
  - Insemine, Porto Alegre, Rio Grande do Sul